CLINICAL TRIAL: NCT00081484
Title: A Randomized, Open-label Study of the Effect of Maintenance Mircera Administered With Pre-filled Syringes on Hemoglobin Levels in Anemic Dialysis Patients With Chronic Kidney Disease
Brief Title: A Study of Intravenous or Subcutaneous Mircera for the Treatment of Anemia in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA17284
Record Dates: First submitted 2004-04-13; First posted 2004-04-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa; continuous erythropoietin receptor activator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- 2 (Active Comparator)
  Interventions: Drug: epoetin alfa or beta

INTERVENTIONS:
Drug: epoetin alfa or beta — iv or sc, as prescribed
  Arms: 2
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 30, 50 or 90 micrograms iv or sc (starting dose) every 2 weeks
  Arms: 1

SUMMARY:
This study will assess the efficacy and safety of intravenous (iv) or subcutaneous (sc) Mircera, administered with pre-filled syringes, as maintenance treatment for renal anemia in chronic kidney disease patients on dialysis who were previously receiving iv or sc epoetin. The anticipated time on study treatment is 3-12 months and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic renal anemia;
* on dialysis therapy for at least 12 weeks before screening;
* receiving iv or sc epoetin for at least 8 weeks before screening.

Exclusion Criteria:

* women who are pregnant, breastfeeding or using unreliable birth control methods;
* administration of another investigational drug within 4 weeks before screening, or during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2004-06; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin concentration | Weeks 1-36

SECONDARY OUTCOMES:
Number of patients maintaining average Hb concentration within +/- 1g/dL of average baseline Hb concentration | Weeks 29-36
RBC transfusions | Weeks 1-36
AEs, laboratory parameters, vital signs | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (61):
- United States (26):
  - Covina, California
  - Los Alamitos, California
  - Los Angeles, California
  - San Diego, California
  - Tampa, Florida
  - Honolulu, Hawaii
  - South Holland, Illinois
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Kalamazoo, Michigan
  - Columbus, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Hackensack, New Jersey
  - Flushing, New York
  - New York, New York
  - Orchard Park, New York
  - Cleveland, Ohio
  - Oregon City, Oregon
  - Erie, Pennsylvania
  - Lewistown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Charlottesville, Virginia
  - Norfolk, Virginia
- Canada (4):
  - Ottawa, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
- France (7):
  - Aix-en-Provence
  - Chambéry
  - Hyères
  - Le Kremlin-Bicêtre
  - Nantes
  - Paris
  - Rouen
- Germany (3):
  - Erlangen
  - München
  - Nuremberg
- Italy (3):
  - Como
  - Modena
  - Pavia
- Poland (2):
  - Rzeszów
  - Warsaw
- Portugal (3):
  - Carnaxide
  - Porto
  - Setúbal
- Puerto Rico (2):
  - Ponce
  - San Juan
- Spain (2):
  - Alicante
  - Madrid
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei
- Bangkok, Thailand
- United Kingdom (5):
  - Glasgow
  - Hertford
  - London
  - Salford
  - Swansea

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280